CLINICAL TRIAL: NCT04220775
Title: Phase I/II Study of M7824 Plus Curative Intent Re-Irradiation With Stereotactic Body Radiation Therapy (SBRT) in Patients With Local-Regionally Recurrent Head and Neck Squamous Cell Carcinoma
Brief Title: Bintrafusp Alfa and Stereotactic Body Radiation Therapy for the Treatment of Recurrent or Second Primary Head and Neck Squamous Cell Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to no longer develop the drug and stop support of studies using the drug.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0608; NCI-2019-07625 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0608 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-26; First posted 2020-01-07 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-07

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma; Second Primary Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — bintrafusp alfa protein, human; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (bintrafusp alfa, SBRT) (Experimental): Patients receive bintrafusp alfa IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Beginning day 15 of cycle 1, patients also undergo SBRT over 5 fractions once QOD for 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bintrafusp Alfa; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Bintrafusp Alfa — Given IV
  Other Names: Anti-PDL1/TGFb Trap MSB0011359C; M7824; MSB0011359C
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I/II trial studies the side effects and how well bintrafusp alfa and stereotactic body radiation therapy work in treating patients with head and neck squamous cell cancer that has come back (recurrent) or has occurred after having cancer in the past (second primary). Immunotherapy with bintrafusp alfa may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving bintrafusp alfa and stereotactic body radiation therapy may help to control recurrent head and neck squamous cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety, tolerability and feasibility of bintrafusp alfa (M7824) when administered together with stereotactic body radiation therapy (SBRT) reirradiation. (Lead In) II. To evaluate the progression-free survival (PFS) rate of M7824 plus SBRT reirradiation at 1 year. (Phase 2)

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate by Response Evaluation Criteria in Solid Tumors (RECIST).

II. To evaluate the 1-year locoregional control (LRC), locoregional failure-free survival (LFFS), distant metastasis (DM) and overall survival (OS) rates.

III. To evaluate acute and late toxicity using Common Terminology Criteria for Adverse Events (CTCAE) - version (v) 5.0.

IV. To evaluate fibrosis-related toxicities and functional outcomes. V. To evaluate patient reported outcome (PRO) measures of symptoms using MD Anderson Symptom Inventory (MDASI).

VI. To evaluate volumetric tumor regression rate and magnetic resonance imaging (MRI) kinetic biomarkers after M7824 plus SBRT.

VII. To compare quality-adjusted-life-years (QALY) between M7824 plus SBRT reirradiation and historic SBRT reirradiation control.

EXPLORATORY OBJECTIVE:

I. Biomarkers will be accessed in the tumor and blood samples and correlated with clinical outcomes and toxicity.

OUTLINE:

Patients receive bintrafusp alfa intravenously (IV) over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Beginning day 15 of cycle 1, patients also undergo SBRT over 5 fractions once every other day (QOD) for 2 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 90 days and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented local-regional recurrent squamous cell carcinoma of the head and neck, or second primary squamous cell carcinoma of the head and neck
* Patients must be willing to undergo research biopsy for tissue collection at baseline and at disease progression
* Previous receipt of at least 30 Gy of radiation for head and neck squamous cell cancer (HNSCC) with overlapping fields
* Not eligible or poor candidate or patient refusal of surgery for recurrence
* Evaluable disease apparent on imaging (MRI or computed tomography [CT])
* 1 to 3 sites of recurrence (< 60 cm^3 per site, total volume < 100 cm^3)
* Eastern Cooperative Oncology Group (ECOG) = 0, 1, or 2
* White blood count (WBC) >= 2000/L
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3
* Platelets >= 100,000 cells/mm^3
* Hemoglobin >= 9.0 g/dl; Note: The use of transfusion or other intervention to achieve hemoglobin (Hgb) >= 9.0 g/dl is acceptable
* Serum creatinine =< 1.5 mg/dl or creatinine clearance (CC) >= 50 ml/min determined by 24-hour collection or estimated by Cockcroft-Gault formula
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (except patients with Gilbert syndrome who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x the upper limit of normal
* Negative serum pregnancy test for women of childbearing potential and confirmation within 24 hours of first dose of study drug

Exclusion Criteria:

* Presence of distant metastases
* Less than six-month disease free interval from end of prior radiotherapy to the head and neck
* Prior receipt of anti-PD-1/L1
* Patients who are pregnant or breast feeding
* Clinically significant uncontrolled major cardiac, respiratory, renal, hepatic, gastrointestinal or hematologic disease but not limited to: symptomatic congestive heart failure, unstable angina, or cardiac dysrhythmia not controlled by pacer device; myocardial infarction within 3 months of registration
* Active autoimmune disorder or immunosuppression (including human immunodeficiency virus [HIV], but excluding endocrine abnormalities that are controlled with replacement medications)
* Active viral hepatitis
* Steroid therapy of greater than prednisone 10 mgs a day or equivalent
* Prior history of invasive non-head and neck cancer within two years, with the exception of screen detected prostate cancer treated with observation only, basal cell and squamous cell carcinoma of the skin, and micro-invasive resected cervical carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrarotto, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Saint A, Van Obberghen-Schilling E. The role of the tumor matrix environment in progression of head and neck cancer. Curr Opin Oncol. 2021 May 1;33(3):168-174. doi: 10.1097/CCO.0000000000000730. PMID 33720067
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 participants were registered, 1 participants were not treated, not eligible or inevaluable, Participant withdrew before screening completed.
Pre-assignment Details: The study was planned to enroll 8 patients in phase 1 to assess safety and toxicity. However, based on sponsored analytical findings of other trials using this drug the sponsor decided to no longer develop the drug and stop support of studies using the drug. The study was ended early. Three participants were registered, 2 of them were treated and 1 of them withdrew before screening completed.
Groups:
- Phase 1 Bintrafusp Alfa + SBRT; Phase 2 Bintrafusp Alfa + SBRT: Participants receive bintrafusp alfa IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Started | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Disease Progression | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 60.4 [40.8 to 80.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: For the phase I part of this phase I/II study, the primary endpoint was DLT defined as any grade 3 or above AE resulting in inability to complete radiotherapy due to toxicity related to M7824 or the combination of M7824 and SBRT.
Time Frame: The DLT window is from first M7824 dose (D0) until 14 days post SBRT (D28).
Population: The two participants who were enrolled in phase 1 part of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 2 | 0
Participants
  DLT | 0 | 0
  No DLT | 2 | 0

2. Secondary Outcome: Progression-free Survival (PFS) Rate at 1 Year
Description: For the phase II part of this phase I/II study, the primary endpoint was to evaluate progression-free survival (PFS) at 1 year. Progression-free survival was defined as from treatment start to progression, or death, whichever occurred first, or to the last follow-up.
Time Frame: Up to 1 year
Population: The study was terminated after enrollment of 2 participants in phase 1 and no participants participated in the phase II part of this study.
Groups:
- Phase 1 Bintrafusp Alfa + SBRT: Patients receive bintrafusp alfa IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Overall Response by RECIST
Description: Best overall response by RECIST 1.1
Time Frame: Tumor reassessment during treatment
Population: The study was terminated after enrollment of 2 patients in phase 1 and no patient participated in the phase II part of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 2 | 0
Participants
  Partial response | 1 | 0
  Progressive disease | 1 | 0

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined was from treatment start to death or to the last follow-up
Time Frame: Up to 1 year
Population: This was a secondary outcome in phase 2 only. The study was terminated after enrollment of 2 patients in phase 1 and no patient participated in the phase 2 part of this study. This outcome was not analyzed because no patient was recruited in phase 2.
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: To Evaluate Acute and Late Toxicity Using Common Terminology Criteria for Adverse Events (CTCAE)-v5.0
Description: Common Terminology Criteria for Adverse Events (CTCAE)-v5.0
Time Frame: Up to 1 year
Population: as for outcome 4
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: To Evaluate Fibrosis-related Toxicities and Functional Outcomes
Time Frame: up to 1 year
Population: as for outcome 4
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: To Evaluate Patient Reported Outcome (PRO) Measures of Symptoms Using MD Anderson Symptom Inventory (MDASI)
Time Frame: up to 1 year
Population: as for outcome 4
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: To Evaluate Volumetric Tumor Regression Rate and MRI Kinetic Biomarkers After M7824 Plus SBRT
Time Frame: up to 1 year
Population: as for outcome 4
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: To Compare Quality-Adjusted-Life-Years (QALY) Between M7824 Plus SBRT Reirradiation and Historic SBRT Reirradiation Control
Time Frame: up to 1 year
Population: as for outcome 4
Arm/Group | Phase 1 Bintrafusp Alfa + SBRT | Phase 2 Bintrafusp Alfa + SBRT
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Bintrafusp Alfa + SBRT: Patients receive bintrafusp alfa IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
Arm/Group | Bintrafusp Alfa + SBRT
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bintrafusp Alfa + SBRT (N=2)
Acute Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bintrafusp Alfa + SBRT (N=2)
Alanine aminotransferase increased (Investigations) | 1 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Investigations - Other, specify (Amylase Increased) (Investigations) | 1 (1)
Investigations - Other, specify (Bilirubin Increased) (Investigations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Osteoarthritis) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Lichen planus of tongue) (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders - Other, specify (N/A) (Nervous system disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Serum amylase increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT04220775/Prot_SAP_000.pdf
  • Informed Consent Form (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/75/NCT04220775/ICF_001.pdf